CLINICAL TRIAL: NCT00261937
Title: Inhaled Furosemide Versus Placebo for Acute Viral Bronchiolitis in Hospitalized Infants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bnai Zion Medical Center (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 67/05
Record Dates: First submitted 2005-12-05; First posted 2005-12-06 (Estimated); Last update posted 2013-02-06 (Estimated); Status verified 2005-12

CONDITIONS: Bronchiolitis
MeSH Terms: conditions — Bronchiolitis | interventions — Saline Solution

INTERVENTIONS:
Drug: Inhaled Furosemide vs Placebo (Normal Saline)

SUMMARY:
We hypothesize that inhaled Furosemide will be an effective treatment in infants with acute bronchiolitis.

ELIGIBILITY:
Inclusion Criteria:

* Age: 0-12 months.
* Infants who are otherwise healthy
* Infants with chronic lung disease of prematurity (BPD) will be included, but will be analyzed separately.
* Parents signed a written informed consent.

Exclusion Criteria:

* • Other previous or co-morbidity, specifically: respiratory (other than BPD, like Asthma or Cystic Fibrosis), cardiac or renal disease or anomaly.

Ages: 1 Day to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 2005-12; Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Clinical respiratory effects

SECONDARY OUTCOMES:
1. The duration of hospitalization
2. Time weaned off oxygen
3. Time to full enteral feeding

CONTACTS AND LOCATIONS:
Overall Officials: Amir Kugelman, Principal Investigator — Bnai Zion Medical Center
Locations (1):
- Bnai Zion Medical Center and Naharia Galilli Medical Center, Haifa, Israel

REFERENCES:
- [Result] Bar A, Srugo I, Amirav I, Tzverling C, Naftali G, Kugelman A. Inhaled furosemide in hospitalized infants with viral bronchiolitis: a randomized, double-blind, placebo-controlled pilot study. Pediatr Pulmonol. 2008 Mar;43(3):261-7. doi: 10.1002/ppul.20765. PMID 18214942